CLINICAL TRIAL: NCT02827578
Title: Efficacy and Safety of Tamsulosin/Solifenacin Combination Therapy in Patients With Voiding Symptoms and Moderate to Severe Storage Symptoms Due to Benign Prostate Hyperplasia : a Randomized, Double Blinded, Parallel Design, Active Controlled, Multi-center, Phase 3 Clinical Trial
Brief Title: Efficacy and Safety of Tamsulosin/Solifenacin Combination Therapy in Patients With Voiding Symptoms and Moderate to Severe Storage Symptoms Due to Benign Prostate Hyperplasia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID-TASO-301
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-04

CONDITIONS: Benign Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tamsulosin + Solifenacin (Experimental): Tamsulosin and Solifenacin
  Interventions: Drug: Tamsulosin; Drug: Solifenacin
- Tamsulosin + Solifenacin Placebo (Active Comparator): Tamsulosin and Solifenacin placebo
  Interventions: Drug: Tamsulosin; Drug: Solifenacin placebo

INTERVENTIONS:
Drug: Tamsulosin — Tamsulosin
Drug: Solifenacin — Solifenacin
  Arms: Tamsulosin + Solifenacin
Drug: Solifenacin placebo — Solifenacin placebo
  Arms: Tamsulosin + Solifenacin Placebo

SUMMARY:
Efficacy and Safety of Tamsulosin/Solifenacin Combination therapy in Patients with voiding symptoms and moderate to severe storage symptoms due to Benign Prostate Hyperplasia : a randomized, double blinded, parallel design, active controlled, multi-center, phase 3 clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male aged 45 years old or older
2. Subjects with benign prostatic hyperplasia diagnosed by digital rectal examination
3. Subjects with lower urinary tract symptom suggestive of benign prostate hyperplasia, who spontaneously agree to join and sign to the consent form

Exclusion Criteria:

1. Subjects who have a history of the lower urinary tract cancer, including prostate cancer and bladder cancer within the past 5 years
2. Subjects who have acute urinary retention within 4 weeks before screening
3. Subjects who have clinically significant severe cardiovascular disease(unstable angina, myocardial infarction or arrhythmia) within 6 months before screening
4. Subjects who have hypersensitivity to investigational product or sulfa medications
5. Subjects who were suspected or confirmed calculus of lower urinary tract, calculus of bladder (except for complete recovery,)
6. Subjects who have myasthenia gravis, narrow angle glaucoma or autonomic neuropathy
7. Subjects who have cataract or glaucoma scheduled to be operated in the study duration.
8. Subjects who have hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
9. Subjects who are judged by the investigators to be unsuitable to participate in the clinical trial.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The change of TUFS((Total Urgency and Frequency Score)/24h | From baseline at week 12
The change of total IPSS(International prostate symptom score) | From baseline at week 12

SECONDARY OUTCOMES:
The change of urgency/24h | From baseline at week 4, 8 and 12
The change of voiding frequency/24h | From baseline at week 4, 8 and 12
The change of nocturnal frequency/24h | From baseline at week 4, 8 and 12
The change of urge urinary incontinence frequency/24h | From baseline at week 4, 8 and 12
The change of IPSS(International prostate symptom score)-sub score | From baseline at week 4, 8 and 12
The change of PPBC(Patient perception of bladder condition) | From baseline at week 4 and 12
The change of IPSS(International prostate symptom score) QoL(Quality of Life) | From baseline at week 4, 8 and 12
PGIC(Patient Global Impression of change) and CGIC(Clinician Global Impression of change) | From baseline at week 12
The ratio of subjects who are decreased total IPPS(International prostate symptom score) more than 4 | From baseline at week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No